CLINICAL TRIAL: NCT05036018
Title: RanDOmized stUdy Comparing Both Latest Generation Self-Expanding Valves and a Minimalist approaCH vs. Standard Of Care In transCathEter Aortic Valve Implantation
Acronym: DOUBLE-CHOICE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Leipzig Heart Science gGmbH (Other)
Collaborators: Heart Center Leipzig - University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0165
Record Dates: First submitted 2021-08-30; First posted 2021-09-05 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Aortic Valve Stenosis
Keywords: TAVI; ACURATE neo2; Evolut Pro; local anesthesia; conscious sedation; monitored anesthesia care; minimalist approach
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Patient Reported Outcome Measures; Standard of Care

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to one of four treatment groups in a 1:1:1:1 ratio
Masking Description: Blinding of cardiologists, anesthesiologists and patients is not possible due to the type of interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Active Comparator): Patients treated with the ACURATE neo2 valve using a minimalist approach
  Interventions: Device: ACURATE neo2; Procedure: minimalist approach
- Group 2 (Active Comparator): Patients treated with the ACURATE neo2 valve under standard of care
  Interventions: Device: ACURATE neo2; Procedure: Standard of care
- Group 3 (Active Comparator): Patients treated with the Evolut Pro, Pro+ or FX valve using a minimalist approach
  Interventions: Procedure: minimalist approach; Device: CoreValve Evolut Pro, Pro+ and FX
- Group 4 (Active Comparator): Patients treated with the Evolut Pro, Pro+ or FX valve under standard of care
  Interventions: Device: CoreValve Evolut Pro, Pro+ and FX; Procedure: Standard of care

INTERVENTIONS:
Device: ACURATE neo2 — The ACURATE neo2 valve will be implanted using a two-step mechanism during transfemoral transcatheter aortic valve implantation (TAVI). Balloon predilatation will be recommended in the ACURATE neo 2 valve group.
  Arms: Group 1; Group 2
Procedure: minimalist approach — Isolated local anesthesia. Central venous lines, additional arterial lines for blood pressure monitoring, and urinary catheters will be avoided. Insertion of temporary pacemakers is optional and should be avoided whenever possible, and peri-procedural pacing can then be performed on the left ventricular wire. Patients will be directly transferred to the cardiology ward after the procedure, which can be postponed in case of complications.
  Arms: Group 1; Group 3
Device: CoreValve Evolut Pro, Pro+ and FX — The Evolut Pro, Pro+ or FX valve is positioned in a controlled manner either without pacing or under 'slow-rapid' pacing with allowance for limited repositioning and is anchored to the annulus and ascending aorta.
  Arms: Group 3; Group 4
Procedure: Standard of care — Sedation should be titrated to a Richmond Agitation Sedation Scale (RASS) of 0 to -2 according to local standard of care.The use of EEG monitoring (i.e. BIS, Sedline) can be applied. Continuous CO2-monitoring via face mask should be established during sedation. All patients will receive supplemental oxygen by face mask to maintain an oxygen saturation of approximately 95%. The use of central venous catheters, additional arterial lines for blood pressure monitoring, and urinary catheters can be implemented according to local institutional standards.
  Arms: Group 2; Group 4

SUMMARY:
Open-label, 2 x 2 factorial, prospective, randomized, national, multicenter study to compare latest-generation self-expanding valves and a minimalist approach versus standard of care in transcatheter aortic valve implantation.

DETAILED DESCRIPTION:
The purpose of the DOUBEL-CHOICE study is to demonstrate non-inferiority of a latest-generation self-expanding valve (SEV) (ACURATE neo2, Boston Scientific, Marlborough, MA, USA) in comparison to another latest-generation SEV (Evolut Pro, Pro+ and FX, Medtronic Inc., Minneapolis, MN, USA) and of a minimalist approach vs. standard of care with respect to safety and efficacy in patients with severe symptomatic aortic stenosis undergoing transfemoral TAVI.

ELIGIBILITY:
Inclusion Criteria:

* Severe symptomatic aortic valve stenosis (AVA ≤1 cm² or 0.6 cm²/m²) with indication for transcatheter aortic valve implantation according to heart team consensus
* Perimeter-derived native aortic valve annulus diameter measuring 21-27 mm
* Heart team consensus that the patient is anatomically suitable for both device types
* Suitability for transfemoral vascular access
* Written informed consent

Exclusion Criteria:

* Life expectancy <12 months due to comorbidities
* Native aortic valve annulus <21 mm and >27 mm
* Bicuspid aortic valve
* Cardiogenic shock or hemodynamic instability
* Active endocarditis
* Contraindications for transfemoral access
* Active peptic ulcer or upper gastro-intestinal bleeding <2 weeks
* Hypersensitivity or contraindication to aspirin, heparin or clopidogrel
* Contraindication for a specific treatment strategy (minimalist approach vs. standard of care) as judged by the Heart Team
* Clear patient-specific clinical or anatomic reasons to prefer one treatment strategy or valve type over the other
* Active infection requiring antibiotic treatment
* Age <18 years
* Participation in another interventional trial where the primary endpoint has not been reached

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 836 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2035-02-01 (Estimated)

PRIMARY OUTCOMES:
Devices: Composite of all-cause mortality, stroke, moderate or severe prosthetic valve regurgitation, and permanent pacemaker implantation at 30-day follow-up | Day 30
Strategy: composite of all-cause mortality vascular complications (major + minor according to VARC-3), bleeding complications (type 1-4 according to VARC-3), infections requiring antibiotic treatment, and neurologic events (NeuroARC type 1-3) | Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Holger Thiele, Prof. Dr., Study Chair — Heart Center Leipzig at University of Leipzig, Department of Internal Medicine/Cardiology
Locations (10):
- Germany (10):
  - Zentralklinik Bad Berka, Bad Berka
  - Herz- und Diabeteszentrum NRW, Bad Oeynhausen
  - Universitätsklinikum Köln, Cologne
  - St.-Johannes-Hospital Dortmund, Dortmund
  - Universitätsklinikum Gießen, Giessen
  - Heart Center Leipzig at University of Leipzig, Department of Internal Medicine/Cardiology, Leipzig
  - Herzzentrum München, München
  - LMU Klinikum München, München
  - Universitätsklinikum Tübingen, Tübingen
  - Helios Klinikum Wuppertal, Wuppertal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Feistritzer HJ, Ender J, Lauten P, Rudolph TK, Rudolph V, Geisler T, Massberg S, Adam M, Baldus S, Sossalla S, Joner M, Mollmann H, Wolf A, Kim WK, Borger MA, Noack T, Magunia H, von Dossow V, Sander M, Vigelius-Rauch U, Feuerecker M, Zakhary W, Boening A, Bleiziffer S, Hohenstein S, Hoesler N, Buske M, Desch S, Abdel-Wahab M, Thiele H; DOUBLE-CHOICE Investigators. Peri-Interventional Anesthesia Strategies for Transcatheter Aortic Valve Implantation: A Multicenter, Randomized, Controlled, Noninferiority Trial. Circulation. 2025 Dec 2;152(22):1526-1537. doi: 10.1161/CIRCULATIONAHA.125.076557. Epub 2025 Aug 29. PMID 40878766